CLINICAL TRIAL: NCT06931860
Title: Comparative Effectiveness of Mailed Cologuard Outreach to Mailed FIT Outreach
Brief Title: Head to Head Trial of Mailed Cologuard to Mailed FIT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joshua Demb, PhD, MPH, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 80312400; R00CA267181 (NIH); 4R00CA267181-03 (NIH)
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer Screening; Fecal Immunochemical Test; Multi-target Stool DNA; Colorectal Cancer (CRC)
Keywords: screening; early detection; colorectal cancer; stool blood test; mailed outreach
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Two-arm intervention trial comparing mailed Cologuard outreach (Intervention 1) to mailed FIT outreach (Intervention 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Mailed Cologuard Outreach (Experimental): Receipt of mailed Cologuard test for colorectal cancer screening to be completed and returned by participant. If test is negative, participant will be advised to undergo another test in 3 years. If test is positive, participant will be advised to schedule colonoscopy for further testing.
  Interventions: Diagnostic Test: Cologuard
- Mailed Fecal immunochemical test Outreach (Experimental): Receipt of mailed FIT for colorectal cancer screening to be completed and returned by participant. If test is negative, participant will be advised to undergo another test in 1 year. If test is positive, participant will be advised to schedule colonoscopy for further testing.
  Interventions: Diagnostic Test: Fecal Immunochemical Test

INTERVENTIONS:
Diagnostic Test: Cologuard — Multi-target stool DNA test for colorectal cancer screening implemented by Exact Sciences. Cologuard has 94% sensitivity and 87% specificity to detect colorectal cancer.
  Arms: Mailed Cologuard Outreach
Diagnostic Test: Fecal Immunochemical Test — Stool blood test for colorectal cancer screening. FIT has 75% sensitivity and 90% specificity to detect colorectal cancer.
  Arms: Mailed Fecal immunochemical test Outreach

SUMMARY:
The objective of this study is to measure the comparative effectiveness of mailed outreach of two stool based tests, multi-target stool DNA (Cologuard) and the fecal immunochemical test (FIT) in screening eligible adults ages 45-49 receiving care at the University of California San Diego Health system.

DETAILED DESCRIPTION:
Adults ages 45-49 who are insured, deemed average risk and not currently up to date with colorectal cancer screening will be enrolled. Eligible participants will be randomized to either mailed Cologuard outreach, facilitated by Exact Sciences or mailed FIT outreach. Colorectal cancer screening completion within 12 months of randomization will be measured as the primary outcome, in addition to secondary outcomes of Cologuard or FIT positivity rate measured within 12 months of randomization, and follow-up colonoscopy uptake and CRC incidence, measured within 24 months of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 45-49 with EHR documentation indicating that the patient has an assigned primary care provider at UCSD Health
* ≥1 UCSD Health System health visit within the last year
* Resides in San Diego or Imperial County
* Currently not up to date with CRC screening
* Insured by private, public or other health insurance.

Exclusion Criteria:

* Up-to-date with screening
* Prior history of colonic disease, including inflammatory bowel disease, one or more colorectal neoplastic polyps (i.e., adenomas) or colorectal cancer.
* Prior history of colectomy
* Lack of health insurance

Ages: 45 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of Colorectal cancer screening completion | Within 12 months of randomization
  The proportion of individuals who complete any colorectal cancer screening test recommended by US Preventive Services Task Force (colonoscopy, FIT, Cologuard, Sigmoidoscopy or CT Colonography)

SECONDARY OUTCOMES:
Proportion of Abnormal stool blood test results | Within 12 months of randomization
  Among those completing designed interventions (Cologuard or FIT), the proportion of test results yielding an abnormal result.
Proportion of Follow-up colonoscopy after abnormal stool blood test result | Within 24 months after randomization
  Among those with positive stool blood test results, the proportion who complete diagnostic follow-up colonoscopy
Colorectal cancer incidence | Within 24 months after randomization
  Number of colorectal cancers detected during study period

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Demb, PhD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Data being used for this project involves protected health information that requires special training and completion of research proposals, IRB applications and data use requests directly with University of California San Diego Health System to obtain access. Therefore, we do not anticipate creating unique data resources as part of this study. If researchers receive permission via IRB applications and data use requests to work with these data, we will make available individual-level scientific data used in our study.
  The rationale is based on restrictions put forth as part of our Institutional Review Board (IRB) protocol and the need to protect study participants from risks associated with their participation. Specifically, our study outlines that data access will be limited to study personnel and will only be accessible for those individuals who have IRB-required training with access to a secure HIPAA research server.